CLINICAL TRIAL: NCT06200415
Title: Glucosamine Sulphate Versus Ginger as an Adjunctive Local Delivery Agents in Non-Surgical Periodontal Therapy (A Randomized Controlled Clinical Trial With Biochemical Analysis)
Brief Title: Glucosamine Sulphate Versus Ginger in Non-Surgical Periodontal Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana Ali Mohamed Ali El-Gohary, Post graduate student, department of Oral Medicine, Periodontology, Oral Diagnosis and Radiology, Faculty of Dentistry, Ain Shams University, Egypt), Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDASU-Rec IM012013
Record Dates: First submitted 2023-12-28; First posted 2024-01-11 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Pocket
Keywords: glucosamine sulphate; ginger; local delivery
MeSH Terms: conditions — Periodontal Pocket | interventions — Glucosamine; ginger extract

STUDY DESIGN:
Intervention Model Description: supra and sub gingival scaling will be performed to all patients followed by application of local delivery drug within two groups to assess the effects after 1 month then 3 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucosamine sulphate gel (Experimental): injecting about 2 mm of glucosamine sulphate gel in the affected periodontal pocket only once
  Interventions: Drug: Glucosamine Sulfate
- ginger gel (Experimental): injecting about 2 mm of ginger gel in the affected periodontal pocket only once
  Interventions: Drug: Ginger Oil

INTERVENTIONS:
Drug: Glucosamine Sulfate — Glucosamine sulphate (GLcN) is an N-deacetyl amino sugar derived from the complete hydrolysis of the chitosan with significant anti-inflammatory action.
  Other Names: Glucosamine sulphate
  Arms: Glucosamine sulphate gel
Drug: Ginger Oil — Ginger (Zingiber officinale Roscoe) has been found to have biological activities such as antioxidant, anti-inflammatory, antimicrobial, and anticancer activities.
  Other Names: Ginger; Zingiber officinale; Zingiber genus
  Arms: ginger gel

SUMMARY:
Glucosamine (GlcN) is an N-deacetyl amino monosaccharide sugar derived from complete hydrolysis of chitosan in which it is important vector for chondroitin and keratin sulfate, while on the other hand, medicinal plants became a source of great economic benefit worldwide, ginger has been found to have biological activities such as antioxidant, anti-inflammatory, antimicrobial, and anticancer activities. So, these effects which made it a good candidate to be used in periodontal therapy. The main objective of this study is to assess and compare the effect of locally delivered glucosamine sulphate gel versus ginger gel on the clinical parameters in periodontitis patients including Plaque index (PI), Means sulcus bleeding index (MSBI), Probing depth (PD), Clinical attachment loss (CAL). and to detect the effect of locally delivered both gels on RANKL level in gingival crevicular fluid.

DETAILED DESCRIPTION:
Periodontitis was described as a chronic multifactorial inflammatory disease associated with formation of plaque biofilms and characterized by progressive destruction of the tooth-supporting apparatus. Its primary manifestation includes the loss of periodontal tissue support, featured through clinical attachment loss (CAL) and radiographically alveolar bone loss with the presence of periodontal pockets which are a significant mark of the disease, hence, can progressively lead to tooth loss and gingival bleeding.

The new classification of periodontal and peri-implant diseases and conditions in 2017 classified these diseases into four main categories: First category concerned with periodontal health & gingival diseases either dental biofilm induced gingivitis or non-dental biofilm induced gingivitis. Second category concerned with periodontitis which can be classified into necrotizing periodontitis, periodontitis as a manifestation of systemic disease and periodontitis which include the forms of the disease previously recognized as "chronic" or "aggressive". Third category concerned with other conditions can affect the periodontium as systemic diseases, traumatic occlusion, mucogingival deformities, tooth related factors, periodontal abscesses and endodontic-periodontal diseases. Fourth category concerned with peri-implant diseases and conditions as peri-implant health, peri-implant mucositis, peri-implantitis and peri-implant soft & hard tissue deficiencies.

But now, Periodontitis can be described into four stages depending on the clinical attachment loss (CAL) starting from Stage 1: Initial periodontitis (CAL 1-2 mm), Stage 2: Moderate periodontitis (CAL 3-4 mm), Stage 3: Severe periodontitis with potential for additional tooth loss and Stage 4: Severe periodontitis with potential for loss of dentition (CAL ≥5 mm). Grading focuses on assessment of the risk factors as smoking, systemic factors as diabetes, and outcomes of non-surgical periodontal therapy. Grade A: Slow rate of progression (no CAL loss over 5 years), Grade B: Moderate rate of progression (CAL loss <2 mm over 5 years) and Grade C: Rapid rate of progression (≥2 mm over 5 years).

The pathogenesis of periodontal diseases is mediated by the inflammatory response to bacteria in the dental biofilm. The immune response to infection is regulated by cytokine and chemokine signals. Cytokines and chemokines (chemotactic cytokines) are the messages between cells. Cytokines are low-molecular-weight proteins involved in the initiation and advanced stages of inflammation, in which they can regulate the amplitude and the duration of the response. The genetic regulation leading to the secretion of proinflammatory cytokines from various cells is generally depending on the activation of nuclear factor kappa-B transcription. Cytokines are produced by resident cells, such as epithelial cells and fibroblasts, and by phagocytes (neutrophils and macrophages) in the acute and early chronic phases of inflammation, and by immune cells (lymphocytes) in early and advanced lesions. After recognition of the presented microbes to the appropriate cells, cytokines of the innate response, including tumor necrosis factor alpha, interleukin-1beta and interleukin-6, are the first to face in the pathogenesis pathways of the periodontal disease. It is suggested that individuals who produce high levels of these mediators in response to such thing will go through more and severe tissue loss.

In General, periodontitis is a chronic inflammation in which elimination of the virulent factors can be necessary in treatment of periodontitis by initial intervention by scaling and root surface debridement So, we should know about the importance of human gingival fibroblasts (HGFs). First, HGFs represent most prominent cells in periodontal tissue. Lipopolysaccharides (LPS)-treated HGFs produce inflammatory cytokines such as IL-6 and IL-8 and inflammatory chemical mediators such as Prostaglandin (PGE2), and second; HGFs continue to produce PGE2 IL-6, and IL-8 in the presence of LPS, unlike macrophages. So, it is known that large number of chemical mediators and cytokines was obtained from HGFs can be within the periodontal tissues. That kind of oral infection can be restricted by using antimicrobial mouth wash such as chlorhexidine. usual handling of these chemicals may induce unwanted adverse effects such as tooth staining, taste alteration and development of hypersensitivity reactions.

Antibiotics such as penicillin have been notified for dental caries prevention in humans and animals, merely they reported many side effects, added to the development of the bacterial resistance, so here comes the reason for a deep need for natural antibacterial substitutes. One of the strongest substitutes are medicinal plants.

Glucosamine is a biological element of joint cartilage, it has been known as popular systemic supplement combined with chondroitin sulfate for knee osteoarthritis (OA), as so these compounds could have a chondro-protective effect on knee OA. It is an amino monosaccharide in which it is important vector for chondroitin and keratin sulfate and also, an independent meta-analysis has shown that in trials using a particular formulation of glucosamine as the crystalline glucosamine sulfate (pCGS) gives better result on pain than other preparations of glucosamine did. Glucosamine has a role as a part of glucosaminoglycans (GAGs), it reveals an anti-inflammatory action in vitro and in vivo GlcN reduce the releasing of inflammatory mediators such as nitric oxide (NO), prostaglandin (PG) E2 and interleukin (IL)-8 by chondrocytes and synovial cells. These outcomes propose that GlcN expresses an anti-inflammatory effect on chondrocytes and synovial cells, hence revealing a protective action on OA. Chondroitin-sulphate (CS) and glycosamine-sulphate (GS) has proved a direct effect on OA in combination or alone, as CS has a direct effect on suppressing the production of osteoprotegerin OPG and RANKL the main two major factors involved in the remodeling process, and GS especially has a significant effect. In vitro studies have shown that glucosamine prevents bone resorption by means of down-regulation of RANKL expression in the joints, through lowering the number of RANKL positive T cells and the level of sRANKL in the joint's extracts.

On the other hand, medicinal plants became a source of great economic benefit worldwide. The recent natural recipes utilizing medicinal plants is giving a natural replacement for antibiotic unpleasant effects such as supra infections, hypersensitivity reaction and teeth staining. In addition, using of systemic antibiotics against oral infections is not recommended because of the risk for development of bacterial resistance. However, the discovery of natural extracts of medicinal plants with antimicrobial and anti-inflammatory activity will be valuable and safe.

Ginger (Zingiber officinale Roscoe), which belongs to the Zingiberaceae family and the Zingiber genus, has been commonly consumed as a spice and an herbal medicine for a long time. Bioactive compounds such as terpene and phenolic compounds have been recognized in ginger. The phenolic compounds are mainly gingerols, shogaol, and paradols, they resemble for different bioactivities of ginger. Ginger has been found to have biological activities such as antioxidant, anti-inflammatory, antimicrobial, and anticancer activities. A lot of studies have revealed that ginger can affect many diseases, such as cardiovascular diseases, neurodegenerative diseases, obesity, diabetes mellitus, chemotherapy-induced nausea and emesis, and respiratory disorders. So, more attention will be focused on the bioactivities of the ginger.

In fresh ginger the major polyphenols are gingerols such as 6-gingerol, 8-gingerol, and 10-gingerol. Which if heat treated or stored for long time turns into into corresponding shogaol and after hydrogenation, shogaol can be transformed into paradols. It was found that overproduction of free radicals, such as reactive oxygen species (ROS), plays a strong role in the initiation of many chronic diseases.

Antioxidant activity: studies have shown that ginger has a protective effect against reactive oxygen species (ROS) as it showed antioxidant effects in the chondrocyte cells of human, with oxidative stress mediated by interleukin-1β (IL-1β). It lowers the production of ROS and lipid peroxidation and stimulates the expression of several antioxidant enzymes (). Ginger and its bioactive compounds (such as 6-shogaol) exerting an antioxidant role via the nuclear factor erythroid 2-related factor 2 (Nrf2) signaling pathway.

Anti-Inflammatory Activity: several studies has conveyed that ginger, and its active compounds has anti-inflammatory activity which can protect against inflammation-related diseases The anti-inflammatory effects were mostly related to phosphatidylinositiol -3-kinase (PI3K), protein kinase B (Akt), and the nuclear factor kappa light chain-enhancer of activated B cells (NF-κB). Adding that 6-shogaol exhibited a protective impact against tumor necrosis factor α (TNF-α). It also down regulates the Claudin-2 and the disassembly of Claudin-1 via the suppression of signaling pathways involved with PI3K/Akt and NF-κB. Moreover, nanoparticles derived from edible ginger (GDNPs 2) could increase the levels of anti-inflammatory cytokines such as interleukin-10 (IL-10) and IL-22 and decreasing the levels of pro-inflammatory cytokines such as TNF-α, IL-6, and IL-1β specifically nanoparticles loaded with 6-shogaol so help in lowering the inflammatory process.

Cytotoxicity: Ginger has been examined and considered for its anticancer properties against different types of cancers, such as breast, cervical, prostate, and colorectal cancer Where its mechanisms of action are represented in the inhibition of proliferation and the induction of apoptosis in cancer cells.

Antidiabetic Activity: Diabetes mellitus is known as a serious metabolic disorder condition caused by insulin deficiency and/or insulin resistance, which results in an abnormal rising in blood glucose. Prolonged hyperglycemia could speed up the protein glycation production which results in formation of advanced glycation end products (AGEs). An in vitro study resulted in both 6-shogaol and 6-gingerol preventing the progression of diabetic complications, and how they prevent the production of AGEs by trapping methyl-glyoxal (MGO), the precursor of AGEs Other several studies have investigated the antidiabetic effect of ginger and its major active elements.

ELIGIBILITY:
Inclusion Criteria:

* Localized periodontitis, probing depth ≥5 mm. Less than 30% of teeth are involved.
* Age ranging from 25 to 50 years.
* Good compliance with the plaque control instructions following initial therapy.
* Availability for follow up and maintenance program.
* Systemically free according to the American Society of Anesthesiologists (ASA I).

Exclusion Criteria:

* Smokers
* Systemic diseases which could influence the outcome of the therapy (According to Cornell Medical Index-Health Questionnaire).
* Pregnant and lactating females.
* Vulnerable groups of patients' e.g. (prisoners, handicapped patients and decision ally impaired individuals).
* Unwilling patients to perform oral hygiene measures of plaque control.
* Patients with a history of allergy against any components of the two materials.
* Previous Periodontal treatment or any use of antibiotic/anti-inflammatory drugs within the last 6 months before the initiation of the study

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Assess the effect of locally delivered glucosamine sulphate gel versus ginger gel on Plaque index PI in periodontitis patients | 1 month and three months
  Assess the effect of locally delivered glucosamine sulphate gel versus ginger gel on Plaque index PI (0-3 score) in periodontitis patients
Assess the effect of locally delivered glucosamine sulphate gel versus ginger gel on Mean Sulcus Bleeding Index MSBI in periodontitis patients | 1 month and three months
  Assess the effect of locally delivered glucosamine sulphate gel versus ginger gel on Mean Sulcus Bleeding Index MSBI (0-5 score) in periodontitis patients
Assess the effect of locally delivered glucosamine sulphate gel versus ginger gel on Probing depth PD in periodontitis patients | 1 month and three months
  Assess the effect of locally delivered glucosamine sulphate gel versus ginger gel on Probing depth PD in millimeters in periodontitis patients
Assess the effect of locally delivered glucosamine sulphate gel versus ginger gel on clinical attachment loss (cal) in periodontitis patients | 1 month and three months
  Assess the effect of locally delivered glucosamine sulphate gel versus ginger gel on clinical attachment loss (cal) in millimeters in periodontitis patients

SECONDARY OUTCOMES:
2. Detect the effect of locally delivered glucosamine sulphate and ginger gels on receptor activator nuclear factor kappa B ligand (RANKL) level in gingival crevicular fluid | 1 month and three months
  2. Detect the effect of locally delivered glucosamine sulphate and ginger gels on receptor activator nuclear factor kappa B ligand (RANKL) level in g/ml in gingival crevicular fluid

CONTACTS AND LOCATIONS:
Overall Officials: Hala A. Abuel Ela, professor, Study Director — Faculty of dentistry- Ain Shams University; Olfat G. Shaker, professor, Study Director — Cairo University; Dina A. Othman, professor, Study Director — Faculty of pharmacy- Azhar University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical effect of subgingivally delivered simvastatin in the treatment of patients with chronic periodontitis: a randomized clinical trial — http://pubmed.ncbi.nlm.nih.gov/20151799/
- See also: Chondroitin and glucosamine sulfate in combination decrease the pro-resorptive properties of human osteoarthritis subchondral bone osteoblasts: a basic science study — http://pubmed.ncbi.nlm.nih.gov/17996099/
- See also: Gingerdione A, a polyphenol present in ginger, suppresses obesity and adipose tissue inflammation in high-fat diet-fed mice — http://pubmed.ncbi.nlm.nih.gov/28556482/
- See also: 6-Paradol and 6-Shogaol, the Pungent Compounds of Ginger, Promote Glucose Utilization in Adipocytes and Myotubes, and 6-Paradol Reduces Blood Glucose in High-Fat Diet-Fed Mice — http://pubmed.ncbi.nlm.nih.gov/28106738/
- See also: Edible ginger-derived nanoparticles: A novel therapeutic approach for the prevention and treatment of inflammatory bowel disease and colitis-associated cancer — http://pubmed.ncbi.nlm.nih.gov/27318094/